CLINICAL TRIAL: NCT03999840
Title: A Phase II, Randomized, Double-blind, Placebo-controlled Trial to Evaluate the Safety and Efficacy of Cemdisiran (ALN-CC5) Following Withdrawal of Chronic Eculizumab Therapy in Patients With Atypical HUS at High Risk of Recurrence
Brief Title: Eculizumab to Cemdisiran Switch in aHUS
Acronym: DANCE
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to the COVID global pandemic Sponsor has not received the economic support necessary for the study conduction.
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Cemdisiran in aHUS; 2018-004382-13 (EudraCT Number)
Record Dates: First submitted 2019-06-25; First posted 2019-06-27 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Atypical Hemolytic Uremic Syndrome
Keywords: aHUS; cemdisiran; synthetic RNA interference
MeSH Terms: conditions — Atypical Hemolytic Uremic Syndrome

STUDY DESIGN:
Intervention Model Description: This will be a prospective, randomized, double blind, placebocontrolled trial organized in a Core Study, an Extension follow-up period and a Safety Period.
  The study duration for each patient is 108 weeks (core study 32 weeks, extension follow up 52 weeks and safety follow up 24 weeks).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In order to have a balanced distribution of risk factors for disease recurrence and considering the small number of patients and of expected events, before randomization patients will be stratified according to previous history of disease relapse (after eculizumab interruption and/or after a course of plasma therapy) YES or NO.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMP (Experimental): Cemdisiran (600 mg) or placebo will be administered subcutaneously every four weeks up to week 32 (end of the Core Study).
  Interventions: Drug: cemdisiran
- Placebo (Placebo Comparator): Cemdisiran (600 mg) or placebo will be administered subcutaneously every four weeks up to week 32 (end of the Core Study).
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: cemdisiran — Cemdisiran has been designed to reduce the level of C5 mRNA in the liver, thereby reducing levels of circulating C5 protein, inhibiting terminal complement pathway activity, and preventing formation and deposition of the MAC (C5-b9) on endothelial cells in the kidney.
  Other Names: ALN-CC5
  Arms: IMP
Drug: Placebos — The control drug for this study will be a placebo (sodium chloride 0.9% w/v for SC administration). Placebo will be prepared and labelled identically to cemdisiran.
  Arms: Placebo

SUMMARY:
Atypical Hemolytic Uremic Syndrome (aHUS) is a rare, lifethreatening, chronic disease of complement-mediated thrombotic microangiopathy (TMA) characterized by acute onset of renal impairment, thrombocytopenia, and microangiopathic hemolytic anemia. The estimated incidence of aHUS is approximately 0.5 per million per year. aHUS affects both adults and children, but is observed primarily in children and young adults.

Atypical HUS commonly develops due to dysregulation of the alternative complement pathway and can be sporadic (80%) or familial(20%).

The clinical course of aHUS is often unpredictable and can be dependent upon the specific genetic abnormality present within the complement system, if any, and/or triggering events associated with complement activation or inflammation, including autoimmune disease, transplant, pregnancy, infection, metabolic conditions, and drug use. In patients with dysregulated complement activity, such as those with complement mutations commonly observed in aHUS, the kidney vasculature is often the site of thrombosis stemming from endothelial injury.

Cemdisiran has been designed to reduce the level of C5 mRNA in the liver, thereby reducing levels of circulating C5 protein, inhibiting terminal complement pathway activity, and preventing formation and deposition of the MAC (C5-b9) on endothelial cells in the kidney. As a result, complement-mediated endothelial cell damage in patients with aHUS and subsequent progression to End Stage Renal Disease (ESRD) may be reduced.

ELIGIBILITY:
Inclusion Criteria:

1. 12 years and older at the time of consent;
2. Written informed consent (of parents or the guardian in case of underage participants) to enter the study;
3. Consent to stop eculizumab therapy during the whole study period and to resume eculizumab therapy in case of disease recurrence
4. >40 kg body weight;
5. On stable disease status with eculizumab continuous therapy for aHUS for ≥ 12 consecutive months (stability assessed on the basis of hematological/biochemical parameters by the Investigator)
6. Hematological remission at screening and inclusion;
7. Estimated GFR (by the simplified MDRD equation) > 30/ml/min 1.73 m2;
8. Known high risk of aHUS recurrence due to at least one of the following criteria;

   1. History of aHUS recurrence after interruption of eculizumab therapy;
   2. Plasma dependent and/or recurrent disease before the introduction of eculizumab therapy;
   3. Documented mutations in complement factors that are associated with a high risk of disease recurrence such as mutations in Factor H, I or B;
9. Females childbearing potential and non-sterile males must agree to use a method of contraception;
10. Documented previous immunisation against Neisseria meningitidis (serotypes A, C, Y, W135 e B) by anti A, C, W and Y vaccine and anti B vaccine (Bexsero®) and antibiotic prophylaxis in accordance with the KDIGO guidelines and local standard of care of the PI at the trial Center, OR de-novo immunisation against Neisseria meningitidis and antibiotic prophylaxis in accordance with the KDIGO guidelines and local standard of care of the PI at the trial Center, if necessary. Documented previous immunization against Streptococcus pneumoniae and Haemophilus influenzae type b (Hib). Study participants who do not have a sufficient history for some or all of these vaccines should be vaccinated.

Exclusion Criteria:

1. Solid organ or bone marrow/stem cell transplantation;
2. Alanine transaminase (ALT) >3×ULN, INR >2 (or >3.5 if on anticoagulants), or total bilirubin >3×ULN (unless bilirubin elevation is due to Gilbert's syndrome);
3. Clinical or biochemical evidence of active thrombotic; microangiopathy or flare of aHUS at the time of enrolment
4. Evidence of Shigatoxin associated HUS;
5. Patients who required intensified eculizumab therapy because of uncontrolled disease (these patients could be at very high risk of relapse after the shift, even in the cemdisiran treatment arm and their inclusion could be unsafe);
6. Patients who did not relapse despite prolonged (>3 months) interruption of eculizumab therapy (these would probably be low risk patients that are expected to be event-free throughout the whole study period independent of treatment allocation and could have a dilution effect for event analyses);
7. Patients with a confirmed diagnosis of sepsis, defined as positive blood cultures within 7 days of the screening visit and not treated with antibiotics to which the organism is sensitive;
8. Presence or suspicion of active and untreated systemic bacterial infection that, in the opinion of the Investigator confounds an accurate diagnosis of aHUS or impedes the ability to manage the aHUS disease;
9. Evidence of human immunodeficiency virus (HIV) (positive serology for HIV antibody [HIV Ab]), hepatitis B infection (positive hepatitis B surface antigen [HbsAg]), or hepatitis C infection (positive anti-HCV antibody [HCV Ab]) at Screening or historically
10. Unresolved meningococcal disease;
11. Known Systemic Lupus Erythematosus (SLE) or antiphospholipid antibody positivity or syndrome;
12. Exposure to any other investigational drug acting directly on the complement system (except for eculizumab) within 5 half-lives of screening is prohibited;
13. Chemotherapeutic agents within 3 months of enrolment in the study are prohibited;
14. History of malignancy within 5 years of screening;
15. Participation in other clinical trials within 4 weeks of signing the consent form;
16. Active systemic autoimmune diseases other than the target condition. Dermatologic diseases such as atopic dermatitis or psoriasis will not be a reason for exclusion unless there are associated systemic symptoms such as arthritis;
17. Any severe systemic disorder that could interfere with the evaluation of the study treatment (e.g. hepatic disease) that in the opinion of the Investigator would affect the outcome of the study or interfere with interpretation of results;
18. Failure to satisfy the Investigator of fitness to participate for any other reason or any condition (e.g. severe depression or psychiatric disorder) that, in the opinion of the Investigator, could increase the subject's risk by participating in the study or confound the outcome of the study;
19. If female, the subject is pregnant or lactating or intending to become pregnant before, during, or within 90 days after last dose; or intending to donate ova during such time period;
20. If male, the subject intends to donate sperm while on the study or for 90 days after last study drug administration;
21. The subject has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within one year prior to screening. Alcohol abuse is defined as regular weekly intake of >14 units (unit: 1 glass of wine [125 mL] =1 measure of spirits=1/2 pint [0.25 mL] of beer). Alcohol is limited to no more than 2 units per day for the duration of the study;
22. Patients with a poor prognosis that is expected to limit their life expectancy to less than 3 months, in the opinion of the Investigator;
23. History of multiple drug allergies or history of allergic reaction to an oligonucleotide or GalNAc;
24. History of intolerance to subcutaneous (SC) injection(s) or significant abdominal scarring that could potentially hinder cemdisiran administration or evaluation of local tolerability.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Ex vivo complement activation on the surface of cultured microvascular endothelial cells exposed to patient sera | Changes from baseline and 16,32,44,60, 84 and 108 weeks after randomization.
  Persistent inhibition of serum-induced complement (C5b-9) deposition on ADP-activated cultured HMEC-1 (deposition <150%: upper limit of normal range) up to week 32 (Core study) during cemdisiran therapy as compared to complement reactivation during placebo treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro di Ricerche Cliniche per le Malattie Rare " Aldo e Cele Daccò", Ranica, BG, Italy

IPD SHARING:
Plan to Share IPD: No